CLINICAL TRIAL: NCT02364765
Title: Assessment of Changes of Hematological Parameters and Need for Blood Transfusion in Bimaxillary Orthognathic Surgery
Brief Title: Assessment of Hematologic Parameters Before and After Bimaxillary Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antônio Luís Neto Custódio, Associate Professor, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0267.0.203.000-10
Record Dates: First submitted 2015-02-04; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Surgical Blood Loss
Keywords: Maxillofacial Orthognathic Surgery; Hemoglobin; Red Blood Cells; Hematocrit; Blood Platelets; Body Weight; Operative Time; Age Groups; Gender
MeSH Terms: conditions — Blood Loss, Surgical; Body Weight; Coitus | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orthognatic surgery (Other): Elective bimaxillary orthognathic surgery consisting of a unsegmented LeFort I osteotomy combined with a bilateral sagittal split osteotomy, under the influence of mean remifentanil administration of 0.3 mg/kg/hour.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Elective bimaxillary orthognathic surgery consisting of a unsegmented LeFort I osteotomy combined with a bilateral sagittal split osteotomy, under the influence of mean remifentanil administration of 0.3 mg/kg/hour
  Other Names: Ultiva

SUMMARY:
The purpose of the present study was to compare some hematologic parameters and operation time in patients who underwent esthetic bimaxillary surgery under hypotensive anesthesia.

DETAILED DESCRIPTION:
Patients who underwent bimaxillary surgery were prospectively evaluated. Patients were divided into groups based on the surgical procedure and sex (predictor variables). Hemoglobin, red blood cells, hematocrit, and platelet were the primary outcome variables, operation time was the secondary outcome variable, and the patients' age and weight were the other variables.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients listed for elective bimaxillary osteotomies for orthognathic correction by one surgical team, and admitted from August 2010 until June 2012.

Exclusion Criteria:

* Patients who were having single maxillary osteotomies, Le Fort II and III osteotomies, those with general contraindications for extensive surgical intervention, syndromic patients, those with cleft palate, and those with general diseases or hematological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in hematologic parameters | From immediately before the surgery until 24 h after operation
  Hemoglobin (g/dL), red blood cells (cells/mcL), hematocrit (volume %), platelet (cells/mcL)

CONTACTS AND LOCATIONS:
Overall Officials: Antônio LN Custódio, DDS MSc PhD, Principal Investigator — Department of Morphology, Institute of Biological Sciences, Federal University of Minas Gerais
Locations (1):
- Department of Oral and Maxillofacial Surgery - Baleia Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Chrcanovic BR, Toledo GL, Amaral MB, Custodio AL. Assessment of hematologic parameters before and after bimaxillary orthognathic surgery. Oral Maxillofac Surg. 2016 Mar;20(1):35-43. doi: 10.1007/s10006-015-0525-2. Epub 2015 Aug 18. PMID 26280080